CLINICAL TRIAL: NCT03217396
Title: Identification of New Biomarkers Useful to Define the Course of Multiple Sclerosis and Study of the Mechanisms That Promote Synaptic Damage
Brief Title: Biomarkers of Synaptic Damage in Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Collaborators: IRCCS Multimedica (Other)
Responsible Party: Principal Investigator, Mario Stampanoni Bassi, Principal Investigator, Neuromed IRCCS
Other Study IDs: IRCCS Neuromed
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis; Parkinson Disease; Amyotrophic Lateral Sclerosis; Alzheimer Disease
Keywords: synaptic plasticity; neuroinflammation; neurodegeneration
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease; Amyotrophic Lateral Sclerosis; Alzheimer Disease; Neuroinflammatory Diseases; Nerve Degeneration | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- multiple sclerosis patients: lumbar puncture, microRNAs quantification in blood and CSF samples, SNPs analysis
  Interventions: Procedure: lumbar puncture
- neurodegenerative disease patients: lumbar puncture, microRNAs quantification in blood and CSF samples, SNPs analysis
  Interventions: Procedure: lumbar puncture
- control subjects: lumbar puncture, microRNAs quantification in blood and CSF samples, SNPs analysis
  Interventions: Procedure: lumbar puncture

INTERVENTIONS:
Procedure: lumbar puncture — lumbar puncture performed to detect OCB for diagnostic purposes

SUMMARY:
A prospective and retrospective cohort study of about five years will be performed on blood and cerebrospinal fluid samples taken for diagnostic reasons from recruited patients within the Neuromed Neurology Unit. Subjects with other chronic neurodegenerative diseases such as Amyotrophic lateral sclerosis (ALS), Alzheimer's disease (AD) and Parkinson's disease (PD), and healthy subjects subjected to blood sampling and / or lumbar puncture for clinical reasons will be recruited As control groups.

DETAILED DESCRIPTION:
Blood and cerebrospinal fluid samples will be subjected to the procedures required for the isolation of the different components immediately after the withdrawal. Subsequently, the levels of microRNAs, cytokines, chemokines, cell growth factors, neuronal damage markers (tau, phosphorylated and truncated tau, neurofilaments) and mitochondrial (lactate) and free d-amino acids (Objective 1) will be determined. Furthermore, synaptic alterations will be evaluated in the ex vivo chimeric model of MS, using the patch-clamp technique (Objective 2). Genotyping studies will be conducted in order to identify single nucleotide polymorphisms (SNPs) in coding and / or regulating regions of genes (microRNAs or proteins) involved in alterations of the synaptic transmission of MS and its murine experimental model (i.e. SLC1A3, NGFB, PDGFA, etc.), which correlate with specific clinical parameters (i.e. EDSS, BREMS, disease progression index, MS type, disease activity, etc.) and with the levels of potential biomarkers identified

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients (age between 18 and 65 years)
2. Diagnosis of MS in accordance with McDonald's (2010 rev) criteria,
3. EDSS between 0 and 5.5 (included),
4. Patients able to provide informed consent to participation in the study

Exclusion Criteria:

1. Inability to provide informed written consent
2. Altered basal blood count
3. Pregnancy or lactation
4. Contraindications for the execution of magnetic resonance imaging with gadolinium
5. Significant clinical conditions in addition to SM or other chronic neurodegenerative diseases including latent viral infections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients recruited within the Neurology Unit, IRCCS Neuromed. Subjects with other chronic neurodegenerative diseases such as Amyotrophic lateral sclerosis (ALS), Alzheimer's disease (AD) and Parkinson's disease (PD), and healthy subjects subjected to blood sampling and / or lumbar puncture for clinical reasons will be recruited as control group.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive biomarkers of SM using an ex vivo chimeric model | September 01 2020
  CSF concentrations of: neurofilaments, beta amyloid, tau protein, inflammatory cytokines and microRNAs

SECONDARY OUTCOMES:
Identification of new therapeutic targets in MS. | September 01 2020
  CSF concentrations of: neurofilaments, beta amyloid, tau protein, inflammatory cytokines and microRNAs

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, MD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mandolesi G, Rizzo FR, Balletta S, Stampanoni Bassi M, Gilio L, Guadalupi L, Nencini M, Moscatelli A, Ryan CP, Licursi V, Dolcetti E, Musella A, Gentile A, Fresegna D, Bullitta S, Caioli S, Vanni V, Sanna K, Bruno A, Buttari F, Castelli C, Presutti C, De Santa F, Finardi A, Furlan R, Centonze D, De Vito F. The microRNA let-7b-5p Is Negatively Associated with Inflammation and Disease Severity in Multiple Sclerosis. Cells. 2021 Feb 5;10(2):330. doi: 10.3390/cells10020330. PMID 33562569